CLINICAL TRIAL: NCT04048291
Title: Efficacy of Brisk Walking on Improving Balance and Gait Performance, and Functional Mobility in Parkinson's Disease - a Randomized Controlled Trial
Brief Title: Efficacy of Brisk Walking in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Margaret Kit Yi Mak, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20180507003
Record Dates: First submitted 2018-10-09; First posted 2019-08-07 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: rehabilitation; exercise; postural balance
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brisk walking and balance training (Experimental): 1. Week1-6: Supervised training in groups of 6-8 participant, once/week, 90 min/session
  2. Week 7-26: Supervised training in groups of 6-8 participant, once/month, 90 min/session
  3. Participants practice own balance exercise and brisk walking 2-3 times/week (to aim at 150 min of moderate intensity of brisk walking per week at 40-60% of heart rate reserve)
  Interventions: Behavioral: Brisk walking and balance training
- Upper limb exercise (Active Comparator): 1. Week1-6: Supervised training in groups of 6-8 participant, once/week, 90 min/session
  2. Week 7-26: Supervised training in groups of 6-8 participant, once/month, 90 min/session
  3. Participants practice own upper limb exercise 2-3 times/week (to aim at 150 min of exercise per week)
  Interventions: Behavioral: Upper limb exercise

INTERVENTIONS:
Behavioral: Brisk walking and balance training — 6 months of combined brisk walking and balance training
  Arms: Brisk walking and balance training
Behavioral: Upper limb exercise — 6 month of hand dexterity training
  Arms: Upper limb exercise

SUMMARY:
Parkinson's disease (PD) is the second most common neuro-degenerative disease in older people. Falls are common among people PD with the incidence rate up to 70% and have strong associations with the severity of the disease, balance impairment, and freezing of gait.The abnormal gait characteristics include reduction in stride length, gait speed and arm swing, and increase in cadence. Gait training, balance training, aerobic training, Tai chi and dance training are common types of physical rehabilitation for PD. Brisk walking is a way of walking with a pace faster than normal, and it can improve dynamic balance for senior men and balance function for chronic stroke clients.

Brisk walking also promotes cardiopulmonary fitness and walking endurance in elderly women, healthy middle-age and older adults, active elderly men and chronic stroke clients. Our previous pilot randomized controlled trial on the effects of a 6-week home-based brisk walking program indicates that it is feasible and safe for the early PD population with improved walking capacity measured by 6-minute walk distance. The positive effects could carry over to 6 weeks after treatment completion. Up-to-date, the short- and long-term effects of brisk walking in improving balance and gait performance, and functional capacity in people with PD have not yet been well investigated. In order to promote their balance and functional capacity in longer term, more sustained training and better exercise adherence may be necessary.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease diagnosed by neurologist with Hoehn & Yahr stage 2 or 3
* Having a 30-meter walking ability

Exclusion Criteria:

* Significant neurological condition (other than Parkinson's disease)
* Musculoskeletal conditions affecting gait, balance or upper limb functions
* Had received deep brain stimulation surgery
* Cognitive impairment with Montreal Cognitive Assessment score <24
* Present with on-off motor fluctuations.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Mini-Balance Evaluation Systems Test (miniBest) total scores | 1 year
  To evaluate dynamic balance in four domains: anticipatory postural adjustments, postural reactions, sensory integration and gait stability. The miniBEST scores range from 0 to 28, with a higher score indicates better dynamic balance.
Six-minute walking test (6MWT) distance | 1 year
  The maximum walking distance covered during a validated six-minute walk test (6MWT) to document participants' aerobic endurance level and walking capacity
Movement Disorder Society Unified Parkinson Disease Rating Scale Part III (MDS-UPDRS-III) score | 1 year
  This score consists of 18 items in 33 questions examining the motor and functional capacity of people with Parkinson's disease by the assessor. Each question will be rated from 0 (normal) to 4 (severe). The MDS-UPDRS-III score ranges from 0 to 132, with higher scores indicating more severe motor and functional impairments

SECONDARY OUTCOMES:
Fast gait speed | 1 year
  The single-task gait speed measured by a 10-meter walking test in a fast pace
Dual-task timed-up-and-go-time | 1 year
  The dual-task gait performance measured by a 3-meter timed up and go test with serial subtraction
Movement Disorder Society Unified Parkinson Disease Rating Scale Part I (MDS-UPDRS-I) score | 1 year
  This score assesses the non-motor aspects of experiences of daily living in people with Parkinson's disease with a total of 13 questions. The score will be administered by assessor asking participants about their behaviors and non-motor symptoms such as cognitive impairment, hallucination, depressive and anxious mood, sleep, pain, urinary and constipation problems, and fatigue etc. Each question will be rated from 0 (normal) to 4 (severe). The MDS-UPDRS-I score ranges from 0 to 52, with higher scores indicating more severe non-motor impairment.
Activities-specific Balance Confidence (ABC) Scale score | 1 year
  The ABC score will be used to measure the participants' perceived level of balance confidence in 16 indoor and outdoor activities. Each activity is rated from 0-100 (0 indicates no confidence and 100 indicates full confidence, total score=1600). The total score is converted into percentage score ranging from 0 to 100%, with a higher ABC score indicating a higher level of balance confidence.
Parkinson Disease Questionnaire-39 (PDQ-39) summary index score | 1 year
  It is a health-related quality-of-life outcome measure that contains 39 self-reported items on eight domains, i.e.: mobility [#1-10], activities of daily living [#11-16], emotional well-being [#17-22], stigma [#23-26], social support [#27-29], cognition [#30-33], communication [#34-36], and body discomfort [#37-39]. The PDQ-39 has been translated into Chinese and validated for local use. Each item is scored on 5-point Likert-type scales ranging from 0 (never), 1 (occasionally), 2 (sometimes), and 3 (often) to 4 (always) based on their perception on the item over the past month. The PDQ-39 total score is 156 and the PDQ-39 summary index is created by summing all eight of the PDQ-39 domains and standardizing the score on a scale of 0-100%. A lower PDQ-39 summary index score reflects a better health-related quality-of-life.
Fall risk | 1 year
  The risk of falling of each group will be determined by the ratio of non-fallers to fallers at treatment completion and 6-month follow-up. A lower risk ratio indicates a lower risk of falling.
Fall rate | 1 year
  The fall rate (times of fall per year per person) of each group at treatment completion and 6-month follow-up will be calculated with the following formula:
  Number of fall events X12 / (Number of months spent to assemble fall data X number of subjects)
  A lower fall rate indicates a better effect on fall reduction.
Injurious fall risk | 1 year
  The risk of injurious falling of each group at treatment completion and 6-month follow-up will be determined by the ratio of injurious non-fallers to injurious fallers. A lower injurious risk ratio indicates a lower risk of injurious falling.
Injurious fall rate | 1 year
  The injurious fall rate (times of injurious fall per year per person) of each group at treatment completion and 6-month follow-up will be calculated with the following formula:
  Number of injurious fall events X12 / (Number of months spent to collect injurious fall data X number of subjects)
  A lower injurious fall rate indicates a better effect on injurious fall reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret K Mak, Ph.D., Principal Investigator — Department of Rehabilitation Sciences,The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Nothing Selected, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloem BR, Grimbergen YA, Cramer M, Willemsen M, Zwinderman AH. Prospective assessment of falls in Parkinson's disease. J Neurol. 2001 Nov;248(11):950-8. doi: 10.1007/s004150170047. PMID 11757958
- [Background] Pickering RM, Grimbergen YA, Rigney U, Ashburn A, Mazibrada G, Wood B, Gray P, Kerr G, Bloem BR. A meta-analysis of six prospective studies of falling in Parkinson's disease. Mov Disord. 2007 Oct 15;22(13):1892-900. doi: 10.1002/mds.21598. PMID 17588236
- [Background] Wood BH, Bilclough JA, Bowron A, Walker RW. Incidence and prediction of falls in Parkinson's disease: a prospective multidisciplinary study. J Neurol Neurosurg Psychiatry. 2002 Jun;72(6):721-5. doi: 10.1136/jnnp.72.6.721. PMID 12023412
- [Background] Grimbergen YA, Munneke M, Bloem BR. Falls in Parkinson's disease. Curr Opin Neurol. 2004 Aug;17(4):405-15. doi: 10.1097/01.wco.0000137530.68867.93. PMID 15247535
- [Background] Morris ME, Iansek R, Matyas TA, Summers JJ. The pathogenesis of gait hypokinesia in Parkinson's disease. Brain. 1994 Oct;117 ( Pt 5):1169-81. doi: 10.1093/brain/117.5.1169. PMID 7953597
- [Background] Ebersbach G, Sojer M, Valldeoriola F, Wissel J, Muller J, Tolosa E, Poewe W. Comparative analysis of gait in Parkinson's disease, cerebellar ataxia and subcortical arteriosclerotic encephalopathy. Brain. 1999 Jul;122 ( Pt 7):1349-55. doi: 10.1093/brain/122.7.1349. PMID 10388800
- [Background] Mak MK, Wong-Yu IS, Shen X, Chung CL. Long-term effects of exercise and physical therapy in people with Parkinson disease. Nat Rev Neurol. 2017 Nov;13(11):689-703. doi: 10.1038/nrneurol.2017.128. Epub 2017 Oct 13. PMID 29027544
- [Background] Tully MA, Cupples ME, Chan WS, McGlade K, Young IS. Brisk walking, fitness, and cardiovascular risk: a randomized controlled trial in primary care. Prev Med. 2005 Aug;41(2):622-8. doi: 10.1016/j.ypmed.2004.11.030. PMID 15917061
- [Background] Paillard T, Lafont C, Costes-Salon MC, Riviere D, Dupui P. Effects of brisk walking on static and dynamic balance, locomotion, body composition, and aerobic capacity in ageing healthy active men. Int J Sports Med. 2004 Oct;25(7):539-46. doi: 10.1055/s-2004-820948. PMID 15459836
- [Background] Batcho CS, Stoquart G, Thonnard JL. Brisk walking can promote functional recovery in chronic stroke patients. J Rehabil Med. 2013 Sep;45(9):854-9. doi: 10.2340/16501977-1211. PMID 23974944
- [Background] Blain H, Jaussent A, Picot MC, Maimoun L, Coste O, Masud T, Bousquet J, Bernard PL. Effect of a 6-Month Brisk Walking Program on Walking Endurance in Sedentary and Physically Deconditioned Women Aged 60 or Older: A Randomized Trial. J Nutr Health Aging. 2017;21(10):1183-1189. doi: 10.1007/s12603-017-0955-7. PMID 29188878
- [Background] Mak M, Chan W, Auyeung M, Chan A, Cheung N, Mok V. Effects of a home-based brisk walking program in improving activity volume and walking capacity in people with Parkinson's disease. Fourth World Parkinson Congress Abstract; September 2016; Portland 2016.
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886